CLINICAL TRIAL: NCT05804708
Title: A Phase 2 Clinical Trial of GH001 in Patients with Postpartum Depression
Brief Title: Phase 2 Clinical Trial of GH001 in Postpartum Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment of this patient population was more challenging than anticipated. The sponsor concluded that a sufficient amount of patients have completed the trial to demonstrate proof of concept in this patient population.
Sponsor: GH Research Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH001-PPD-203
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Depression; Postnatal Depression
Keywords: Depression; Postpartum Depression; 5-Methoxy-N,N-Dimethyltryptamine; 5-MeO-DMT; Mebufotenin; Postnatal Depression
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GH001 Individualized Dosing Regimen (Experimental): Drug: 5-Methoxy-N,N-Dimethyltryptamine
  GH001 is administered via inhalation, as an IDR (individualized dosing regimen) consisting of up to 3 increasing doses of GH001 (6 mg, 12 mg, and 18 mg), on a single day. The second and third doses are only administered if the patient did not achieve intense psychoactive effects (a peak experience [PE]) at the previously administered dose
  Interventions: Drug: GH001

INTERVENTIONS:
Drug: GH001 — GH001 is administered via inhalation
  Other Names: 5-Methoxy-N,N-Dimethyltryptamine; 5-MeO-DMT; Mebufotenin

SUMMARY:
This study is a multicenter, open-label, single-arm Phase 2 clinical trial. Approximately 15 female participants with clinically diagnosed postpartum depression (PPD) will be included in this study. The participants will receive an individualized dosing regimen (IDR) with at least one and up to three doses of GH001 administered within a single day.

ELIGIBILITY:
Inclusion Criteria:

* Is female and in the age range between 18 and 45 years (inclusive) at screening.
* Has a body mass index (BMI) in the range of 18.5 and 35 kg/m2 (inclusive) at screening.
* Meets the trial criteria for PPD as assessed by a trial psychiatrist or registered clinical psychologist.

Exclusion Criteria:

* Has one or more first or second degree relatives with a current or prior diagnosis of bipolar disorder, psychotic disorder or other mood disorder (including MDD) with psychotic features.
* Current pregnancy resulting in termination, still-birth, pre-term delivery (before week complete gestational week 37), need for intensive care therapy of mother or child, or adoption of child away from patient.
* Has taken prohibited medication or prohibited dietary supplements within the specified timeframe prior to dosing.
* Has previously experienced a significant adverse reaction to a hallucinogenic or psychedelic drug according to the investigator's judgment.
* Has a clinically significant abnormality in physical examination, vital signs, ECG, or clinical laboratory parameters which renders the patient unsuitable for the trial according to the investigator's judgment.
* Patient who has a positive pregnancy test at screening or on the pretest day, is pregnant, or plans to become pregnant during the course of the trial and up to 90 days after GH001 dosing.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
The anti-depressive effects of GH001 evaluated by the change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) assessed at Day 7 | From Baseline to Day 7
  The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. A higher MADRS score indicates more severe depression, and each item is scored from 0 to 6. The overall score ranges from 0 to 60

CONTACTS AND LOCATIONS:
Locations (4):
- Amsterdam UMC, Amsterdam, Netherlands
- United Kingdom (3):
  - Clerkenwell Health, London
  - St. Pancras Clinical Research, London
  - Sheffield Health and Social Care NHS Foundation, Sheffield

IPD SHARING:
Plan to Share IPD: No